CLINICAL TRIAL: NCT04617028
Title: A Randomized, Double-blind, Double-simulated, Parallel-controlled, Multicenter Phase III Study Evaluating the Efficacy and Safety of Jaktinib Versus Hydroxycarbamide in Patients With Intermediate-2 or High-risk Myelofibrosis
Brief Title: Jaktinib Versus Hydroxycarbamide in Subjects With Intermediate-2 or High-risk Myelofibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK016
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib (Experimental): Participants will receive Jaktinib plus placebo to match Hydroxycarbamide.
  Interventions: Drug: Jaktinib; Drug: Placebo to match Hydroxycarbamide
- Hydroxycarbamide (Active Comparator): Participants will receive Hydroxycarbamide plus placebo to match Jaktinib.
  Interventions: Drug: Hydroxycarbamide Tablets; Drug: Placebo to match Jaktinib

INTERVENTIONS:
Drug: Jaktinib — Jaktinib Hydrochloride Tablets administered orally twice daily
  Arms: Jaktinib
Drug: Placebo to match Hydroxycarbamide — Placebo to match Hydroxycarbamide Tablets administered orally twice daily
  Arms: Jaktinib
Drug: Hydroxycarbamide Tablets — Hydroxycarbamide Tablets administered orally twice daily
  Arms: Hydroxycarbamide
Drug: Placebo to match Jaktinib — Placebo to match Jaktinib Tablets administered orally twice daily
  Arms: Hydroxycarbamide

SUMMARY:
This study is to determine the efficacy of Jaktinib versus Hydroxycarbamid in participants with Intermediate-2 or High-risk myelofibrosis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,either male or female;
* Subjects diagnosed with a PMF according to World Health Organiztion criteria (2016 Edition), or patients diagnosed with a Post-PV-MF or Post-EF-MF according to International Working Group for Myeloproliferative Neoplasms Research and Treatment criteria;
* High risk or intermediate-2 risk as defined by the Dynamic International Prognostic Scoring System (DIPSS) for Primary Myelofibrosis;
* Subjects have no plan for stem cell transplantation in the near future;
* Life expectancy of > 24 weeks;
* ECOG performance status of 0-1;
* Palpable splenomegaly at least 5 cm below left costal margin;
* Peripheral blood blast count ≤ 10%;
* Subjects who have not yet received treatment with a JAK inhibitor, or Subjects who have been treated with JAK inhibitors for ≤10 days;
* Subjects have not received growth factor, thrombopoietin mimetics or platelet transfusion(s) within 2 weeks before the randomization; ANC≥ 1.0×10^9/L, platelet count ≥ 100×10^9/L within 2 days before the randomization;
* Normal functions in major organs within 7 days before the randomization, fulfilling the following criteria: ALT and AST ≤ 2.5×ULN; DBIL and TBIL ≤ 2.0×ULN; serum creatinine ≤ 1.5×ULN;
* If the subject is receiving any anti-myelofibrosis treatment (except for JAK inhibitors and hydroxyurea) at screening, the dosing regimen must remain unchanged for at least 2 weeks before screening. If the investigator judges that there is no need to continue to use, stop the use of thalidomide, androgens and prednisone> 10 mg during screening. The drugs used to improve anemia should be stopped for at least 6 half-lives or 2 weeks before randomization(whichever is the longer);
* If the subject is receiving Hydroxycarbamide treatment at screening, the drug must be discontinued ≥ 2 weeks before the randomization;
* Meet the requirements of the ethics committee and willing to sign the informed consent form;
* Ability to comply with trial and follow-up procedures.

Exclusion Criteria:

* Subjects with any significant clinical and laboratory abnormalities which may affect the safety evaluation, such as uncontrolled diabetes, uncontrolled hypertension after taking two or more hypotensive drugs, peripheral neuropathy;
* Subjects with congestive heart failure, uncontrolled or unstable angina or myocardial infarction, cerebrovascular accident, or pulmonary embolism within 24 weeks prior to screening;
* Subjects who have not fully recovered from surgical operation within 4 weeks prior to screening;
* Subjects suffering from arrhythmia and requiring treatment at screening;
* Subjects with clinical symptoms of active bacterial, viral, parasitic or fungal infections requiring treatment at screening;
* Chest X-rays suggest an active lung infection at screening;
* Subjects who had active tuberculosis infection within 48 weeks before screening;γ-Interferon release test suggests latent tuberculosis infection at screening;
* Subjects who had undergone splenectomy, or received radiotherapy to the spleen within 48 weeks before screening;
* Subjects with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC);
* Subjects with epilepsy or patients who have received psychotropic drug or sedatives during screening;
* Female subjects who are pregnant, currently breastfeeding, planning to become pregnant;Subjects who are unable to adopt effective contraceptive methods during the study; Male subjects who did not use condoms during the dosing period and within 2 days after the last dose
* Subjects who had experienced malignant tumors within the past 5 years (except for adequately treated local basal cell carcinoma of the skin and cervical carcinoma in situ that have been cured);
* Subjects who are unsuitable to the trial in combination with other serious diseases, as identified by the investigator;
* Subjects with suspected allergies to Jaktinib or its excipient;
* Subjects who have participated in another clinical trial of a new drug or medical instrument within 12 weeks before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Splenic response rate at Week 24 | Week 24
  Splenic response rate at Week 24 is defined as the proportion of participants achieving a ≥ 35% reduction in spleen volume at Week 24 from baseline as measured by MRI or CT

SECONDARY OUTCOMES:
Proportion of transfusion dependent patients converted to non-transfusion dependent patients at baseline | From start of drug administration up to 7 days after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, PhD, Principal Investigator — The First Affiliated Hospital of Medical School of Zhejiang University
Locations (1):
- The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Zhou H, Suo S, Zhuang J, Yang L, He A, Liu Q, Du X, Gao S, Li Y, Li Y, Chen Y, Wu W, Zhu H, He G, Hong M, Jiang Q, Jiang Z, Jing H, Wang J, Xu N, Yue L, Zheng C, Zhou Z, Jin C, Li X, Liu L, Xu Y, Wu D, Zhang F, Zhang J, Wu L, Yin H, Lv B, Xiao Z, Jin J. Evaluation of gecacitinib vs hydroxyurea in patients with intermediate-2 or high-risk myelofibrosis: final analysis results from a randomized phase 3 study. Blood Cancer J. 2024 Dec 18;14(1):216. doi: 10.1038/s41408-024-01202-8. PMID 39695117